CLINICAL TRIAL: NCT06053424
Title: A Phase 1b Open Label Positron Emission Tomography Study to Assess Changes in Abdominal [11C]AZ14132516 Uptake Following Administration of Single and Repeat Doses of AZD7798 to Healthy Participants and Patients With Crohn's Disease
Brief Title: Positron Emission Tomography (PET) Study of Changes in [11C]AZ14132516 Uptake Following Administration of AZD7798 to Healthy Participants and Patients With Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9690C00004
Record Dates: First submitted 2023-08-30; First posted 2023-09-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Panel 1 (Experimental): Healthy participants will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by a single IV infusion of AZD7798 Dose Level 1 on Day 1. Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 14 and Day 42.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516
- Panel 2 (Experimental): Healthy participants will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by a single IV infusion of AZD7798 Dose Level 2 on Day 1. Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 14 and Day 56.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516
- Panel 3 (Experimental): Healthy participants will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by a single IV infusion of AZD7798 Dose Level 2 on Day 1. Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 2 and Day 42.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516
- Panel 4 (Experimental): Participants with Crohn's disease will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by a single IV infusion of AZD7798 Dose Level 1 on Day 1. Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 14 and Day 42.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516
- Panel 5 (Experimental): Participants with Crohn's disease will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by a single IV infusion of AZD7798 Dose Level 2 on Day 1. Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 14 and Day 42.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516
- Panel 6 (Experimental): Participants with Crohn's disease will receive a single IV bolus dose of radioligand [11^C]AZ14132516 between Day -7 to Day -1 followed by IV infusion of AZD7798 Dose Level 1 on Day 1 (Dose 1) and Day 15 (Dose 2). Thereafter, again will receive IV bolus dose of radioligand [11^C]AZ14132516 on Day 14 and Day 28.
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516

INTERVENTIONS:
Drug: AZD7798 — Participants will receive IV infusion of AZD7798 as stated in arm description.
Drug: [11C]AZ14132516 — Participants will receive IV bolus dose of radioligand [11^C]AZ14132516 as stated in arm description.

SUMMARY:
The purpose of this study is to measure the changes in small bowel uptake of radioligand [11^C]AZ14132516 after intravenous (IV) administration of single and repeat doses of AZD7798 in healthy participants and participants with Crohn's disease.

Study details include:

* The study duration will be variable (adaptive design).
* For Panels 1-5, there will be 5 in-person study visits: 1 screening visit, 1 visit for the baseline PET examination, 1 residential (24 hour) visit for AZD7798 administration and 2 visits for repeated PET examinations. There will be a final follow-up virtual visit (telephone call).
* For Panel 6, there will be 7 in-person study visits: 1 screening visit, 1 visit for the baseline PET examination, 2 residential (24 hour) visits for AZD7798 administration, 1 visit for pharmacokinetic (PK) blood sample and 2 visits for repeated PET examinations. There will be a final follow-up virtual visit.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY PARTICIPANTS:

1. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
2. Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.
3. Participant must be ≥ 20 to 65 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
4. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory parameters, and cardiac monitoring before first administration of investigational product.

   Weight
5. Body weight within 50.0 to 120.0 kg and body mass index within the range 18.0 to 35.0 kg/m^2 (inclusive).
6. Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   1. Male participants:

      * Non-sterilized male participants who are sexually active with a female partner of childbearing potential must use a condom with spermicide during the study period and for at least 7 days following last radioligand administration and 4 months following last dose of AZD7798, whichever is longer.
      * It is strongly recommended that female partners of male participants also use at least one highly effective method of contraception throughout this period.
      * Male participants must refrain from fathering a child or donating sperm during the study period and for at least 7 days following last radioligand administration and 4 months following last dose of AZD7798, whichever is longer.
   2. Female participants:

   (i) Women of non-child bearing potential are defined as meeting one of the following criteria at screening:
   * Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle-stimulating hormone levels in the postmenopausal range.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.

   (ii) Woman of childbearing potential (WOCBP ie, not meeting criteria above) must have a negative pregnancy test at screening and before PET examination.

   (iii) If sexually active with a non-sterilized male partner, WOCBP must use at least one highly effective method of birth control during the study period and for at least 7 days following last radioligand administration and 4 months following last dose of AZD7798, whichever is longer.

   (iv) It is strongly recommended that non-sterilized male partners of WOCBP participants use a male condom plus spermicide during the study period.

   (v) WOCBP participants must not breastfeed and must not donate or retrieve ova for their own use during the study period and for at least 7 days following last radioligand administration and 4 months following last dose of AZD7798, whichever is longer (c) Highly effective methods of birth control (i) Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include:
   * Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
   * Progesterone-only contraception associated with inhibition of ovulation (oral, injectable or implantable)
   * Intrauterine device or hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner (only acceptable if the partner is the sole sexual partner of the participant and the vasectomized partner has received medical assessment of surgical success)
   * Sexual abstinence as defined by refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. It is only acceptable if the preferred and usual lifestyle of the participant.

   PARTICIPANTS WITH CROHN'S DISEASE

<!-- -->

1. As for Healthy Participants (inclusion criteria #1) procedures.
2. Participant must be ≥ 20 to 65 years of age inclusive, at the time of signing the informed consent.
3. Participants with confirmed Crohn's disease with small bowel involvement per study gastroenterologist (diagnosed via combination of clinical findings and at least one of endoscopy and/or histology and/or imaging) with diagnosis made at least 3 months prior to screening.
4. Body weight within 50.0 to 120.0 kg and body mass index within the range 18.0 to 35.0 kg/m^2 (inclusive).
5. As for Healthy Participants (inclusion criteria #6).

Exclusion Criteria:

HEALTHY PARTICIPANTS:

1. Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, hematological disease, hepatic disease, renal disease, gastrointestinal disease, or other major disease.
2. History of cancer with the following exceptions

   (a) Solid malignancy with curative therapy completed at least 5 years prior to screening (b) Basal cell carcinoma or localized squamous cell carcinoma of the skin or in-situ carcinoma of the cervix, provided that curative therapy was completed at least 12 months prior to screening
3. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to biologic therapies.
4. Participants with unstable hypertension (as judged by the Investigator) or symptomatic hypotension, history of pre-syncope or syncope due to orthostatic hypotension and/or induced by change of posture (orthostatic hypotension defined as 25 mmHg decrease in systolic and/or 15 mmHg).
5. Significant abnormalities on clinical examination, including neurological and physical examination, vital signs and electrocardiogram (ECG).
6. Chemistry, hematology, or urine analysis results that may interfere with the study or present a safety risk to the participant.
7. Leukocyte, lymphocyte, or neutrophil counts below the lower limit of normal. A re-test is allowed during screening in cases of mild leukopenia clinically suspected to be transient.
8. Abnormal vital signs, after 10 minutes of supine rest as judged by the investigator. As a guide, any readings outside the following should be considered in the evaluation:

   (a) systolic blood pressure (BP) ≥ 150 mmHg (b) diastolic BP ≥ 90 mmHg (c) heart rate ≤ 35 beats per minute (bpm) or ≥ 100 bpm The inclusion of participants meeting the above criteria may be decided on a case-by case basis by the Principal Investigator (PI).
9. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This may include participants with any of the following:

   1. PR (PQ) interval prolongation of clinical significance as judged by the Investigator
   2. Intermittent second or third-degree atrioventricular (AV) block (AV block II Mobitz type 1, Wenchebach, while asleep or in deep rest is not disqualifying)
   3. Incomplete, full, or intermittent bundle branch block (QRS ≤ 110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy)
   4. Abnormal T wave morphology
   5. Prolonged QTcF ≥ 470 ms or shortened QTcF ≤ 340 ms or a family history of long QT syndrome The inclusion of participants meeting the above criteria may be decided on a case-by case basis by the PI.
10. Positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) serology as defined by:

    (a) Hepatitis B surface antigen (HBsAg) or anti-hepatitis B core antibodies (anti-HBc Ab) positivity (b) Anti-hepatitis C virus antibodies (anti-HCV Ab) positivity (c) Anti-HIV antibodies (Ab) positivity Prior/Concomitant Therapy
11. Participants must abstain from taking prescription or non-prescription drugs (including vitamins, recreational drugs, and dietary or herbal supplements) within 7 days or 5 half-lives (whichever is longer) before the start of study intervention until completion of the follow-up visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
12. Current drug abuse or dependence or positive screen for drugs of abuse at screening visit.
13. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
14. Suffers from claustrophobia that limits the ability to undergo the scanning procedure.
15. Positive Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) rapid antigen test at screening.
16. Any other reason that, in the study PI opinion, prohibits the inclusion of the participants into the study.
17. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
18. Live or attenuated vaccine within 4 weeks of Screening and until the end of the follow-up period and until 12 weeks after the end of the follow-up period (1 year for Bacillus Calmette-Guerin [BCG] vaccination).
19. An active infection, or history of serious infection within the preceding 28 days.
20. Use of antibiotics within 28 days prior to the first administration of investigational medicinal product (IMP), unless, in the opinion of the investigator, the medication will not interfere with the study.
21. History of symptomatic herpes simplex (excluding cold sores) or herpes zoster infection within 3 months prior to screening.
22. Positive or indeterminate tuberculosis (TB) QuantiFERON test.
23. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days/5 half-lives, whichever is longer, of the first administration of IMP in this study. The period of exclusion begins 30 days/5 half-lives, whichever is longer, after the final dose.
24. Participation in a PET imaging research study within last year.

PARTICIPANTS WITH CROHN'S DISEASE

1. Current diagnosis of ulcerative colitis, indeterminate colitis, inflammatory bowel disease unclassified, infectious colitis, or ischemic colitis.
2. History of cytomegalovirus colitis within 12 months prior to screening.
3. Complications of Crohn's Disease including short bowel syndrome, strictures/stenoses with symptomatic obstruction or pre-stenotic dilation, or other conditions where surgery may be anticipated during the study period.
4. Planned bowel or perianal surgery for Crohn's disease prior to end of study follow up visit.
5. Recent bowel resection surgery within 6 months of screening.
6. Participants with undrained fistula or abscess, including active perianal disease.
7. Positive Clostridium difficile toxin test during screening.
8. Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, hematological disease, hepatic disease, renal disease, gastrointestinal disease, or other major diseases other than active Crohn's disease.
9. History of cancer with the following exceptions (a) Solid malignancy with curative therapy completed at least 5 years prior to screening (b) Basal cell carcinoma or localized squamous cell carcinoma of the skin or in-situ carcinoma of the cervix, provided that curative therapy was completed at least 12 months prior to screening
10. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to biologic therapies.
11. Participants with unstable hypertension (as judged by the Investigator) or symptomatic hypotension, history of pre-syncope or syncope due to orthostatic hypotension and/or induced by change of posture (orthostatic hypotension defined as 25 mmHg decrease in systolic and/or 15 mmHg).
12. Significant abnormalities on clinical examination, including neurological and physical examination, vital signs and ECG other than signs of Crohn's disease.
13. Chemistry, hematology, or urine analysis results that may interfere with the study or present a safety risk to the participant.
14. Abnormal vital signs, after 10 minutes of supine rest as judged by the investigator. As a guide, any readings outside the following should be considered in the evaluation:

    1. systolic BP ≥ 150 mmHg
    2. diastolic BP ≥ 90 mmHg
    3. heart rate ≤ 35 bpm or ≥100 bpm The inclusion of participants meeting the above criteria may be decided on a case-by case basis by the PI.
15. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This may include participants with any of the following:

    1. PR (PQ) interval prolongation of clinical significance as judged by the Investigator
    2. Intermittent second or third-degree AV block (AV block II Mobitz type 1, Wenchebach, while asleep or in deep rest is not disqualifying)
    3. Incomplete, full, or intermittent bundle branch block (QRS ≤ 110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy)
    4. Abnormal T wave morphology
    5. Prolonged QTcF ≥ 470 ms or shortened QTcF ≤ 340 ms or a family history of long QT syndrome.

    The inclusion of participants meeting the above criteria may be decided on a case-by case basis by the PI.
16. Positive hepatitis B, hepatitis C or HIV serology as defined by:

    1. HBsAg or anti-HBc Ab positivity
    2. Anti-HCV Ab positivity and HCV RNA positivity
    3. Anti-HIV Ab positivity Prior/Concomitant Therapy
17. Treatment with an anti-tumor necrosis factor (anti-TNF) biologic within 8 weeks of first dose and throughout the study period, unless therapeutic drug monitoring is performed and drug concentrations are undetectable.
18. Treatment with any biologic, other than an anti-TNF (including vedolizumab and ustekinumab) within 12 weeks prior to first dose and throughout the study period, unless therapeutic drug monitoring is performed and drug concentrations are undetectable.
19. Treatment with rituximab within 12 months prior to first dose and throughout the study period.
20. Treatment with Sphingosine-1-phosphate receptor modulators within 12 weeks prior to first dose and throughout the study period.
21. Treatment with Janus Kinase inhibitors within 2 weeks prior to first dose and throughout the study period
22. Treatment with apheresis (eg, Adacolumn, Cellsorba) within 2 weeks prior to first dose and throughout the study period.
23. Treatment with corticosteroids at a total daily dose of greater than 20 mg prednisone or equivalent.
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
25. Suffers from claustrophobia that limits the ability to undergo the scanning procedure.
26. Positive SARS-CoV-2 rapid antigen test at screening.
27. Any other reason that, in the study PI opinion, prohibits the inclusion of the participants into the study.
28. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
29. Live or attenuated vaccine within 4 weeks of screening and until 12 weeks after the end of the follow-up period (1 year for BCG vaccination).
30. An active infection, or history of serious infection within the preceding 28 days.
31. History of symptomatic herpes simplex (excluding cold sores) or herpes zoster infection within 3 months prior to screening.
32. Positive or indeterminate TB QuantiFERON test performed within 1 year of screening (without known interval exposure to TB) or during screening period unless evidence of completion of full treatment course for latent TB with no clinical symptoms or signs indicative of re-activation.
33. Chest x-ray with signs of malignancy or latent or active TB infection performed within 1 year of screening (without known interval exposure to TB) or during screening period.
34. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days/5 half-lives, whichever is longer, of the first administration of IMP in this study. The period of exclusion begins 30 days/5 half-lives, whichever is longer, after the final dose.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Small Bowel Partition Coefficient (Kp) From Baseline (Positron Emission Tomography [PET]1 Visit) to PET2 Visit | PET1 visit (baseline; Day -7 to Day -1) and PET2 visit (Day 14 for all panels except Day 2 for Panel 3)
  Kp is the partition coefficient that denotes radioactivity concentration ratio (area under the concentration-time curve [AUC] 0-60 min, intestines/AUC 0-60 min, blood). Kp denotes that denominator is the radioactivity measurement in blood (aorta), this is the reference region used in calculations. Percentage change in small bowel Kp from baseline (PET1 Visit) to PET2 visit is reported.
Percentage Change in Small Bowel Kp From Baseline (PET1 Visit) to PET3 Visit | PET1 visit (baseline; Day -7 to Day -1) and PET3 visit (Day 42 for all panels except Days 56 and 28 for Panels 2 and 6, respectively)
  Kp is the partition coefficient that denotes radioactivity concentration ratio (area under the concentration-time curve [AUC] 0-60 min, intestines/AUC 0-60 min, blood). Kp denotes that denominator is the radioactivity measurement in blood (aorta), this is the reference region used in calculations. Percentage change in small bowel Kp from baseline (PET1 Visit) to PET3 visit is reported.

SECONDARY OUTCOMES:
Percentage Change From Baseline in Circulating C-C Chemokine Receptor Type 9 Positive (CCR9+) Memory T Cells in Panels 1 to 5 | Panels 1-5: Pre-dose (baseline) and 6 and 24 hours post-dose on Day 1, additionally; Panels 1, 4, and 5: Days 14 and 42; Panel 2: Day 14; Panel 3: Days 2 and 42
  CCR9+ memory T cells in blood were evaluated by flow cytometry. Percentage change from baseline in circulating CCR9+ memory T cells is reported.
Percentage Change From Baseline in Circulating CCR9+ Memory T Cells in Panel 6 | Pre-dose of Dose 1 (baseline), and 6 and 24 hours post-dose 1 on Day 1; pre-dose and 24 hours post-dose 2 on Day 15; and on Day 28
  CCR9+ memory T cells in blood were evaluated by flow cytometry. Percentage change from baseline in circulating CCR9+ memory T cells is reported.
Change From Baseline in C-C Chemokine Receptor Type 9 (CCR9) Receptor Occupancy as Free CCR9 on Total CCR9 Memory T cells in Blood in Panels 1 to 5 | Panels 1-5: Pre-dose (baseline) and 6 and 24 hours post-dose on Day 1, additionally; Panels 1, 4, and 5: Days 14 and 42; Panel 2: Day 14; Panel 3: Days 2 and 42
  CCR9 receptor occupancy as free CCR9 on total CCR9 memory T cells in blood was evaluated by flow cytometry. Change from baseline in CCR9 receptor occupancy as free CCR9 on total CCR9 memory T cells in blood is reported.
Change From Baseline in CCR9 Receptor Occupancy as Free CCR9 on Total CCR9 Memory T cells in Blood in Panel 6 | Pre-dose of Dose 1 (baseline), and 6 and 24 hours post-dose 1 on Day 1; pre-dose and 24 hours post-dose 2 on Day 15; and on Day 28
  CCR9 receptor occupancy as free CCR9 on total CCR9 memory T cells in blood was evaluated by flow cytometry. Change from baseline in CCR9 receptor occupancy as free CCR9 on total CCR9 memory T cells in blood is reported.
Serum Concentrations of AZD7798 in Panels 1 to 5 | Panels 1-5: Pre-dose, 1, 6, 24 hours post-dose on Day 1; additionally, Panels 1, 2, 4, and 5: Day 14; Panel 3: Day 2
  Serum concentrations of AZD7798 collected over time are reported.
Serum Concentrations of AZD7798 in Panel 6 | Pre-dose, 1, 6, and 24 hours post-dose 1 on Day 1; pre-dose, 1, 6, and 24 hours post-dose 2 on Day 15; and on Day 29
  Serum concentration of AZD7798 collected over time are reported.
Maximum Serum Concentration (Cmax) of AZD7798 in Panels 1 to 5 | Panels 1-5: Pre-dose, 1, 6, 24 hours post-dose on Day 1; additionally, Panels 1, 2, 4, and 5: Day 14; Panel 3: Day 2
  The Cmax of AZD7798 is reported.
Cmax of AZD7798 in Panel 6 | Pre-dose, 1, 6, and 24 hours post-dose 1 on Day 1; pre-dose, 1, 6, and 24 hours post-dose 2 on Day 15; and on Day 29
  The Cmax of AZD7798 is reported.
Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Measured Concentration (AUClast) of AZD7798 in Panels 1 to 5 | Panels 1-5: Pre-dose, 1, 6, 24 hours post-dose on Day 1; additionally, Panels 1, 2, 4, and 5: Day 14; Panel 3: Day 2
  The AUClast of AZD7798 is reported.
AUClast of AZD7798 in Panel 6 | Pre-dose, 1, 6, and 24 hours post-dose 1 on Day 1; pre-dose, 1, 6, and 24 hours post-dose 2 on Day 15; and on Day 29
  The AUClast of AZD7798 is reported.
Time to Maximum Serum Concentration (Tmax) of AZD7798 in Panels 1 to 5 | Panels 1-5: Pre-dose, 1, 6, 24 hours post-dose on Day 1; additionally, Panels 1, 2, 4, and 5: Day 14; Panel 3: Day 2
  The Tmax of AZD7798 is reported.
Tmax of AZD7798 in Panel 6 | Pre-dose, 1, 6, and 24 hours post-dose 1 on Day 1; pre-dose, 1, 6, and 24 hours post-dose 2 on Day 15; and on Day 29
  The Tmax of AZD7798 is reported.
Last Measured Serum Concentration (Tlast) of AZD7798 in Panels 1 to 5 | Panels 1-5: Pre-dose, 1, 6, 24 hours post-dose on Day 1; additionally, Panels 1, 2, 4, and 5: Day 14; Panel 3: Day 2
  The Tlast of AZD7798 is reported.
Tlast of AZD779 in Panel 6 | Pre-dose, 1, 6, and 24 hours post-dose 1 on Day 1; pre-dose, 1, 6, and 24 hours post-dose 2 on Day 15; and on Day 29
  The Tlast of AZD7798 is reported.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day -7 to Day -1 through Day 49 for all panels except Panel 2 (Day -7 to Day -1 through Day 63) and Panel 6 (Day -7 to Day -1 through Day 35)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Vital Signs Reported as TEAEs | Day -7 to Day -1 through Day 49 for all panels except Panel 2 (Day -7 to Day -1 through Day 63) and Panel 6 (Day -7 to Day -1 through Day 35)
  Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body temperature, blood pressure, pulse rate, and oxygen saturation).
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs | Day -7 to Day -1 through Day 49 for all panels except Panel 2 (Day -7 to Day -1 through Day 63) and Panel 6 (Day -7 to Day -1 through Day 35)
  Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of clinical chemistry, hematology, coagulation, urinalysis, and drug abuse (healthy participants only).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Creignou, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Research Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/